

**IRAS ID:** 333898

**Study Title:** SOOTH-ED: Purrble's Soothing Touch for Eating Disorders and Autism

## **CONSENT FORM**

| Participant Identification Number: | | |
|---|---|---|
| · | of Researcher: | |
| | | Please<br>initial box |
| 1 | I confirm that I understand that by initialling each box I am consenting to this element of the study. I understand that it will be assumed that uninitialed boxes mean that I DO NOT consent to that part of the study. I understand that by not giving consent for any one element I may be deemed ineligible for the study. | |
| 2 | I confirm that I have read the Participant Information Sheet dated (version 2, 07/02/2024) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | |
| 3 | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | |
| 4 | I consent to the processing of my personal information for the purposes explained to me in the Participant Information Sheet. I understand that such information will be handled in accordance with the terms of the General Data Protection Regulation. | |
| 5 | I consent to receive the questionaries and Purrble Toy (Device under investigation) and agree to complete questionaries and interact with purrble as part of the study. | |
| 6 | I understand that confidentiality and anonymity will be maintained, and it will not be possible to identify me in any research outputs. | |
| 7 | I consent to the direct use of my anonymized quotes in research publications. | |



| | of Person | Date | Signature | <u> </u> |
|---|---|---|---|---|
| Name of Participant | | Date | Signature | |
| * | other research in the | e future and may be sha<br>note that this is optiona | bout me will be used to support<br>red anonymously with other<br>l; you can still participate in the | |
| 9 | I agree to take part i | n the above study. | | |
| | give permission for | where it is relevant to m | ny taking part in this research. I | |
| | the study, may be looked at by individuals from King's College London, from regulatory authorities or | | | |
| 8 | I understand that rel during | evant sections of my me | edical notes and data collected | |

One copy for participant; one copy for study file; one copy for medical notes.